CLINICAL TRIAL: NCT00441259
Title: Randomised, Double Blind, Controlled, Safety, Tolerability and Immunogenicity Phase II Trial of ChimeriVax™-JE and Japanese Encephalitis Inactivated Mouse Brain Vaccine in Children of Descending Age.
Brief Title: Safety and Efficacy Study of ChimeriVax™-JE and JE Inactivated Mouse Brain Vaccine in Children of Descending Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-040-004
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-07

CONDITIONS: Japanese Encephalitis
Keywords: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JE-CV Group (Experimental): Participants will receive Japanese encephalitis chimeric virus vaccine (JE-CV)
  Interventions: Biological: ChimeriVax™-JE
- MBDV Group (Active Comparator): Participants will receive the mouse brain-derived vaccine (MBDV)
  Interventions: Biological: Japanese Encephalitis Inactivated Mouse Brain Vaccine

INTERVENTIONS:
Biological: ChimeriVax™-JE — One dose of 4.0 log10 PFU is given in a volume of 1 ml for children aged > 3 years and 0.5 ml to children and infants aged < 3 years administered subcutaneously
  Arms: JE-CV Group
Biological: Japanese Encephalitis Inactivated Mouse Brain Vaccine — Two doses of 1 ml reconstituted JE-MBDV is given to subjects aged > 3 years and 0.5 ml is given to children and infants aged < 3 years administered subcutaneously
  Arms: MBDV Group

SUMMARY:
This randomised, double-blind study is to be conducted on 96 subjects at multiple sites in India. Subjects will be enrolled by age group and randomised to either ChimeriVax™-JE (JE-CV) or JE Mouse Brain Derived Vaccine (JE-MBDV). Study consists of a screening period, a treatment period and a 2 year follow-up period.

Primary safety endpoints will be the adverse event (AE) rates 28 days after completion of vaccination course. The primary efficacy endpoints will be the rate of seroconversion 28 days after completing vaccination.

ELIGIBILITY:
Inclusion Criteria:

* All aspects of the Protocol explained and written informed consent obtained from the subject's parent or guardian and assent from the child if ≥ 8 years of age.
* Aged ≥ 9 months to < 10 years
* In good general health, without significant medical history, physical examination findings, or clinically significant abnormal laboratory results
* Subject had to be available for the study duration for the study duration, including all planned follow-up visits.

Exclusion Criteria:

* A history of vaccination against, or infection with, JE or other flaviviruses (e.g. Kyanasur Forest Disease, West Nile virus, dengue fever). Previous JE vaccination was to be determined by history (interview of subject's parent or guardian) or by inspecting the child's official vaccination record.
* Demonstration of parasitemia on malaria blood smear at Screening.
* History of residence in or travel to a JE-endemic region of India or elsewhere in Asia (for periods of 4 weeks or more).
* hypersensitivity to thimerosal or gelatin
* Have received a transfusion of blood, blood products or serum globulin in the preceding 6 months,
* Have an immunodeficiency or neurological disorder, or take drugs that suppress the immune system,
* Have a history of severe reaction to other vaccines,
* Have a chronic condition requiring medication,
* Intend to travel out of the area during the study period,
* Have spent at least 4 weeks in a JE-endemic region,
* Plan to receive any other vaccination within the double-blind treatment period, or who have received a vaccination in the month preceding Screening,
* Exhibit signs of secondary or tertiary malnutrition,
* Are seropositive to human immunodeficiency virus (HIV), Hepatitis B or C,
* Have malaria infection, or who have a fever within 3 days before vaccination.
* Those with an acute fever, or with previously scheduled vaccinations, may be rescheduled.
* Consideration of the routine immunisation schedule should be made such that it is ensured that routine vaccinations due are either given before entry to the trial, or afterwards if delayed because of the trial.

Ages: 9 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2007-01; Primary Completion 2011-02 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Dubey, M.D, Principal Investigator — Maulana Azad Medical College, New Delhi, India; Bakul B. Javadekar, M.D., Principal Investigator — Government Medical College, Baroda, India; Atul Shanker, Dr., Principal Investigator — Dr Atul's Child Hospital, Jaipur, Rajasthan, India
Locations (3):
- India (3):
  - Dr Atul's Child Hospital, Jaipur, Rajasthan
  - Government Medical College, Baroda
  - Maulana Azad Medical College, New Delhi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and vaccinated from 03 January 2007 to 13 January 2009 at 3 clinical centers in India.
Pre-assignment Details: A total of 96 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- ChimeriVax™-JE: Participants received one dose of placebo on Day 0 followed by one dose of Japanese encephalitis chimeric virus vaccine (ChimeriVax™-JE) on Day 14.
- Mouse Brain Derived Vaccine: Participants received 2 doses of Japanese encephalitis inactivated mouse brain derived vaccine: 1 dose on Day 0 and 1 dose on Day 14.
Period: Overall Study
Arm/Group | ChimeriVax™-JE | Mouse Brain Derived Vaccine
Started | 48 | 48
Completed | 48 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ChimeriVax™-JE | Mouse Brain Derived Vaccine | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48 | 48 | 96
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 3.8 (2.98) | 3.7 (2.89) | 3.7 (2.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 48
  Male | 21 | 27 | 48
Region of Enrollment [Number; unit: Participants]
  India | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events Following Vaccination With Either ChimeriVax™ JE or JE Inactivated Mouse Brain Derived Vaccine
Time Frame: Day 14 up to Day 42 Post-vaccination
Population: Adverse events were assessed in all enrolled participants, intent-to-treat (safety) population.
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE | Mouse Brain Derived Vaccine
Number analyzed (Participants) | 48 | 48
Participants
  Nasopharyngitis (All; N = 48, 48) | 2 | 2 [0 to 0]
  Otitis Media Acute (All; N = 48, 48) | 1 | 0 [0 to 0]
  Diarrhea Infectious (All; N = 48, 48) | 1 | 0 [0 to 0]
  Dysentery (All; N = 48, 48) | 1 | 0 [0 to 0]
  Hepatitis A (All; N = 48, 48) | 1 | 0 [0 to 0]
  Rash Pustular (All; N = 48, 48) | 1 | 0 [0 to 0]
  Tonsillitis (All; N = 48, 48) | 1 | 0 [0 to 0]
  Upper Respiratory Tract Infection (All; N=48, 48) | 1 | 0 [0 to 0]
  Varicella (All; N = 48, 48) | 1 | 0 [0 to 0]
  Impetigo (All; N = 48, 48) | 0 | 1 [0 to 0]
  Pharyngitis (All; N = 48, 48) | 0 | 1 [0 to 0]
  Viral Upper Respiratory Tract Infect. (All;N=48,48 | 0 | 1 [0 to 0]
  Diarrhea (All; N = 48, 48) | 3 | 2 [0 to 0]
  Vomiting (All; N = 48, 48) | 2 | 1 [0 to 0]
  Haematochezia (All; N = 48, 48) | 1 | 0 [0 to 0]
  Mucous Stools (All; N = 48, 48) | 1 | 0 [0 to 0]
  Constipation (All; N = 48, 48) | 0 | 1 [0 to 0]
  Rhinorrhea (All; N = 48, 48) | 3 | 3 [0 to 0]
  Cough (All; N = 48, 48) | 2 | 2 [0 to 0]
  Wheezing (All; N = 48, 48) | 0 | 2 [0 to 0]
  Pyrexia (All; N = 48, 48) | 2 | 1 [0 to 0]
  Face Edema (All; N = 48, 48) | 1 | 0 [0 to 0]
  Injection Site Pain (All; N = 48, 48) | 1 | 2 [0 to 0]
  Injection Site Swelling (All; N = 48, 48) | 0 | 1 [0 to 0]
  Malaise (All; N = 48, 48) | 1 | 1 [0 to 0]
  Pain (All; N = 48, 48) | 1 | 0 [0 to 0]
  Irritability (All; N = 48, 48) | 0 | 2 [0 to 0]
  Anorexia (All; N = 48, 48) | 2 | 1 [0 to 0]
  Anemia (All; N = 48, 48) | 2 | 2 [0 to 0]
  Eosinophilia (All; N = 48, 48) | 0 | 1 [0 to 0]
  Lacrimation Increased (All; N = 48, 48) | 0 | 1 [0 to 0]
  Laziness (All; N = 48, 48) | 2 | 1 [0 to 0]
  Erythema (All; N = 48, 48) | 1 | 0 [0 to 0]
  Rash (All; N = 48, 48) | 1 | 0 [0 to 0]
  Injury (All; N = 48, 48) | 1 | 0 [0 to 0]
  Eosinophil Count Increased (All; N = 48, 48) | 0 | 1 [0 to 0]
  Hemoglobin Decreased (All; N = 48, 48) | 1 | 0 [0 to 0]
  Pyrexia (≥5 to <10 yr; N = 16, 16) | 2 | 0 [0 to 0]
  Injection Site Pain (≥5 to <10 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Pain (≥5 to <10 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Upper Respiratory Tract Infection (≥5 to <10 yr; | 1 | 0 [0 to 0]
  Eosinophil Count Increased (≥5 to <10 yr; N=16, 16 | 0 | 1 [0 to 0]
  Otitis Media Acute (≥2 to <5 yr: N=16, 16) | 1 | 0 [0 to 0]
  Diarrhea Infectious (≥2 to <5 yr: N=16, 16) | 1 | 0 [0 to 0]
  Hepatitis A (≥2 to <5 yr: N=16, 16) | 1 | 0 [0 to 0]
  Rash Pustular (≥2 to <5 yr: N=16, 16) | 1 | 0 [0 to 0]
  Tonsillitis (≥2 to <5 yr: N=16, 16) | 1 | 0 [0 to 0]
  Varicella (≥2 to <5 yr: N=16, 16) | 1 | 0 [0 to 0]
  Vomiting (≥2 to <5 yr: N=16, 16) | 1 | 0 [0 to 0]
  Injection Site Pain (≥2 to <5 yr: N=16, 16) | 0 | 1 [0 to 0]
  Injection Site Swelling (≥2 to <5 yr: N=16, 16) | 0 | 1 [0 to 0]
  Pyrexia (≥2 to <5 yr: N=16, 16) | 0 | 1 [0 to 0]
  Rhinorrhea (≥2 to <5 yr: N=16, 16) | 1 | 0 [0 to 0]
  Diarrhea (≥9 mo to <2 yr; N = 16, 16) | 3 | 2 [0 to 0]
  Vomiting (≥9 mo to <2 yr; N = 16, 16) | 1 | 1 [0 to 0]
  Haematochezia (≥9 mo to <2 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Mucous Stools (≥9 mo to <2 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Constipation (≥9 mo to <2 yr; N = 16, 16) | 0 | 1 [0 to 0]
  Cough (≥9 mo to <2 yr; N = 16, 16) | 2 | 2 [0 to 0]
  Rhinorrhea (≥9 mo to <2 yr; N = 16, 16) | 2 | 3 [0 to 0]
  Wheezing (≥9 mo to <2 yr; N = 16, 16) | 0 | 2 [0 to 0]
  Nasopharyngitis (≥9 mo to <2 yr; N = 16, 16) | 2 | 2 [0 to 0]
  Dysentery (≥9 mo to <2 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Impetigo (≥9 mo to <2 yr; N = 16, 16) | 0 | 1 [0 to 0]
  Pharyngitis (≥9 mo to <2 yr; N = 16, 16) | 0 | 1 [0 to 0]
  Viral Upper Respiratory Tract Inf (≥9 mo to <2 yr) | 0 | 1 [0 to 0]
  Anorexia (≥9 mo to <2 yr; N = 16, 16) | 2 | 1 [0 to 0]
  Anemia (≥9 mo to <2 yr; N = 16, 16) | 2 | 2 [0 to 0]
  Eosinophilia (≥9 mo to <2 yr; N = 16, 16) | 0 | 1 [0 to 0]
  Irritability (≥9 mo to <2 yr; N = 16, 16) | 0 | 2 [0 to 0]
  Face Edema (≥9 mo to <2 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Malaise (≥9 mo to <2 yr; N = 16, 16) | 1 | 1 [0 to 0]
  Injection Site Pain (≥9 mo to <2 yr; N = 16, 16) | 0 | 1 [0 to 0]
  Laziness (≥9 mo to <2 yr; N = 16, 16) | 2 | 1 [0 to 0]
  Lacrimation Increased (≥9 mo to <2 yr; N = 16, 16) | 0 | 1 [0 to 0]
  Erythema (≥9 mo to <2 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Rash (≥9 mo to <2 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Injury (≥9 mo to <2 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Hemoglobin Decreased (≥9 mo to <2 yr; N = 16, 16) | 1 | 0 [0 to 0]

2. Primary Outcome: Number of Participants With Treatment-Related Adverse Events Following Vaccination With Either ChimeriVax™ JE or JE Inactivated Mouse Brain Derived Vaccine
Time Frame: Day 14 up to Day 42 Post-vaccination
Population: Adverse events were assessed all enrolled and vaccinated participants, intent-to-treat (safety) population.
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE | Mouse Brain Derived Vaccine
Number analyzed (Participants) | 48 | 48
Participants
  Nasopharyngitis (All; N = 48, 48) | 2 | 2 [0 to 0]
  Upper Respiratory Tract Infection (All; N =48, 48) | 1 | 0 [0 to 0]
  Impetigo (All; N = 48, 48) | 0 | 1 [0 to 0]
  Pharyngitis (All; N = 48, 48) | 0 | 1 [0 to 0]
  Diarrhea (All; N = 48, 48) | 1 | 2 [0 to 0]
  Vomiting (All; N = 48, 48) | 1 | 1 [0 to 0]
  Hematochezia (All; N = 48, 48) | 1 | 0 [0 to 0]
  Mucous Stools (All; N = 48, 48) | 1 | 0 [0 to 0]
  Rhinorrhea (All; N = 48, 48) | 1 | 3 [0 to 0]
  Cough (All; N = 48, 48) | 2 | 2 [0 to 0]
  Wheezing (All; N = 48, 48) | 0 | 2 [0 to 0]
  Pyrexia (All; N = 48, 48) | 2 | 0 [0 to 0]
  Injection Site Pain (All; N = 48, 48) | 1 | 2 [0 to 0]
  Injection Site Swelling (All; N = 48, 48) | 0 | 1 [0 to 0]
  Malaise (All; N = 48, 48) | 1 | 0 [0 to 0]
  Pain (All; N = 48, 48) | 1 | 0 [0 to 0]
  Irritability (All; N = 48, 48) | 0 | 1 [0 to 0]
  Anorexia (All; N = 48, 48) | 1 | 1 [0 to 0]
  Anemia (All; N = 48, 48) | 1 | 0 [0 to 0]
  Lacrimation Increased (All; N = 48, 48) | 0 | 1 [0 to 0]
  Rash (All; N = 48, 48) | 1 | 0 [0 to 0]
  Pyrexia (≥5 to <10 yr; N = 16, 16) | 2 | 0 [0 to 0]
  Injection Site Pain (≥5 to <10 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Pain (≥5 to <10 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Upper Respiratory Tract Infection (≥5 to <10 yr) | 1 | 0 [0 to 0]
  Injection Site Pain (≥2 to <5 yr; N = 16, 16) | 0 | 1 [0 to 0]
  Injection Site Swelling (≥2 to <5 yr; N = 16, 16) | 0 | 1 [0 to 0]
  Diarrhea (≥9 mo to <2 yr; N = 16, 16) | 1 | 2 [0 to 0]
  Vomiting (≥9 mo to <2 yr; N = 16, 16) | 1 | 1 [0 to 0]
  Hematochezia (≥9 mo to <2 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Mucous Stools (≥9 mo to <2 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Cough (≥9 mo to <2 yr; N = 16, 16) | 2 | 2 [0 to 0]
  Rhinorrhea(≥9 mo to <2 yr; N = 16, 16) | 1 | 3 [0 to 0]
  Wheezing (≥9 mo to <2 yr; N = 16, 16) | 0 | 2 [0 to 0]
  Nasopharyngitis (≥9 mo to <2 yr; N = 16, 16) | 2 | 2 [0 to 0]
  Impetigo (≥9 mo to <2 yr; N = 16, 16) | 0 | 1 [0 to 0]
  Pharyngitis (≥9 mo to <2 yr; N = 16, 16) | 0 | 1 [0 to 0]
  Anorexia (≥9 mo to <2 yr; N = 16, 16) | 1 | 1 [0 to 0]
  Anemia (≥9 mo to <2 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Irritability (≥9 mo to <2 yr; N = 16, 16) | 0 | 1 [0 to 0]
  Malaise (≥9 mo to <2 yr; N = 16, 16) | 1 | 0 [0 to 0]
  Injection Site Pain (≥9 mo to <2 yr; N = 16, 16) | 0 | 1 [0 to 0]
  Lacrimation Increased (≥9 mo to <2 yr; N = 16, 16) | 0 | 1 [0 to 0]
  Rash (≥9 mo to <2 yr; N = 16, 16) | 1 | 0 [0 to 0]

3. Primary Outcome: Number of Participants With Seroconversion After Vaccination With Either ChimeriVax™ JE or JE Inactivated Mouse Brain Derived Vaccine
Description: Antibodies to Japanese encephalitis (JE) virus were measured with 50% plaque reduction neutralization tests (PRNT50) using JE CV virus, JE virus Nakayama strain, and JE virus strain 826309 (Indian wild-type). Seroconversion was defined as a titer ≥10 1/dil for participants who were seronegative at baseline and ≥ 4 fold rise for participants who were seropositive at baseline (titer ≥ 10 1/dil).
Time Frame: Day 42 Post-vaccination
Population: Seroconversion was assessed all participants who received all doses of the investigational product in the Treatment Period, had Baseline and post-vaccination samples (Day 42) for antibody analysis, per-protocol population.
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE | Mouse Brain Derived Vaccine
Number analyzed (Participants) | 33 | 35
Participants
  Homologous JE-CV virus PRNT (N = 33, 0) | 33 | NA [0 to 0] — Homologous JE-CV virus PRNT used for the assessment of the immune response in ChimeriVax™-JE Vaccine recipients only
  Homologous virus Nakayama strain PRNT (N = 0, 35) | NA — Homologous virus Nakayama strain used for the assessment of the immune response in Mouse Brain Derived Vaccine recipients only | 8
  JE-CV PRNT (N = 33, 35) | 33 | 33 [0 to 0]
  Nakayama PRNT (N = 32, 35) | 8 | 8 [0 to 0]
  Indian WT virus PRNT (N = 33, 35) | 27 | 26 [0 to 0]

4. Primary Outcome: Geometric Mean Titers (GMTs) of Japanese Encephalitis Viruses After Vaccination With Either ChimeriVax™ JE or JE Inactivated Mouse Brain Derived Vaccine
Description: Antibodies to Japanese encephalitis (JE) virus were measured with 50% plaque reduction neutralization tests (PRNT50) using JE CV virus, JE virus Nakayama strain, and JE virus strain 826309 (Indian wild-type).
Time Frame: Day 42 Post Dose 1
Population: Geometric Mean Titers were assessed in participants who received all doses of the investigational product in the Treatment Period, had Baseline and post-vaccination blood samples (Day 42) for antibody analysis, per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ChimeriVax™-JE | Mouse Brain Derived Vaccine
Number analyzed (Participants) | 34 | 35
Titers
  Homologous JE-CV virus PRNT (N = 34, 0) | 313.5 [40 to 5120] | NA [NA to NA] — Homologous JE-CV virus PRNT used for the assessment of the immune response in ChimeriVax™-JE Vaccine recipients only
  Homologous virus Nakayama strain PRNT (N = 0, 35) | NA [NA to NA] — Homologous virus Nakayama strain used for the assessment of the immune response in Mouse Brain Derived Vaccine recipients. | 8.0 [5 to 160]
  JE-CV PRNT (N = 34, 35) | 313.5 [40 to 5120] | 49.7 [5 to 320]
  Nakayama PRNT (N = 33, 35) | 7.8 [5 to 160] | 8.0 [5 to 160]
  Indian WT virus PRNT (N = 34, 35) | 60.1 [5 to 2560] | 17.1 [5 to 320]

5. Secondary Outcome: Number of Participants With Seroconversion After Vaccination With Either ChimeriVax™ JE or JE Inactivated Mouse Brain Derived Vaccine
Description: as for outcome 3
Time Frame: Day 42 Post Dose 1
Population: Seroprotection was assessed in participants who received all doses of the investigational product in the Treatment Period, had Baseline and post-vaccination blood samples (Day 42) for antibody analysis, per-protocol population.
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE | Mouse Brain Derived Vaccine
Number analyzed (Participants) | 34 | 35
Participants
  Homologous JE-CV virus PRNT (N = 33, 0) | 33 | NA [0 to 0] — Homologous JE-CV virus PRNT used for the assessment of the immune response in ChimeriVax™-JE Vaccine recipients only
  Homologous virus Nakayama strain PRNT (N=0,35) | NA — Homologous virus Nakayama strain used for the assessment of the immune response in Mouse Brain Derived Vaccine recipients | 8
  JE-CV Virus (All; N = 33, 35) | 33 | 33 [0 to 0]
  Nakayama Strain (All; N = 32, 35) | 8 | 8 [0 to 0]
  Wild Type Virus (All; N = 33, 35) | 27 | 26 [0 to 0]
  JE-CV Virus (≥5 to <10 yr; N = 12, 13) | 12 | 12 [0 to 0]
  JE Virus Nakayama strain (≥5 to <10 yr; N =12, 13) | 6 | 0 [0 to 0]
  Wild Type Virus (≥5 to <10 yr; N = 12, 13) | 12 | 11 [0 to 0]
  JE-CV Virus (≥2 to <5 yr; N = 8, 9) | 8 | 9 [0 to 0]
  JE Virus Nakayama strain (≥2 to <5 yr; N = 9, 9) | 1 | 6 [0 to 0]
  Wild Type Virus (≥2 to <5 yr; N = 8, 9) | 2 | 6 [0 to 0]
  JE-CV Virus (≥9 mo to <2 yr; N = 13, 13) | 13 | 12 [0 to 0]
  JE Virus Nakayama (≥9 mo to <2 yr; N = 11, 13) | 1 | 2 [0 to 0]
  Wild Type Virus (≥9 mo to <2 yr; N=13, 13) | 13 | 9 [0 to 0]

6. Secondary Outcome: Geometric Mean Titers (GMTs) Using Neutralizing Antibody to Japanese Encephalitis Viruses After Vaccination With Either ChimeriVax™ JE or JE Inactivated Mouse Brain Derived Vaccine
Description: as for outcome 4
Time Frame: Day 42 Post-vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ChimeriVax™-JE | Mouse Brain Derived Vaccine
Number analyzed (Participants) | 34 | 35
Titers
  JE-CV Virus (All; N = 34, 35) | 313.5 [40 to 5120] | 49.7 [5 to 320]
  JE Nakayama Strain (All; N = 33, 35) | 7.8 [5 to 160] | 8.0 [5 to 160]
  Wild Type Virus (All; N = 34, 35) | 60.1 [5 to 2560] | 17.1 [5 to 320]
  JE-CV Virus (≥5 to <10 yr; N = 12, 13) | 226.3 [80 to 5120] | 34.1 [5 to 160]
  JE Virus Nakayama Strain (≥5 to <10 yr; N =12, 13) | 13.3 [5 to 160] | 5.0 [5 to 5]
  Wild Type virus (≥5 to <10 yr; N = 12, 13) | 100.8 [10 to 2560] | 17.0 [5 to 40]
  JE-CV Virus (≥2 to <5 yr; N = 9, 9) | 254.0 [80 to 1280] | 74.1 [40 to 160]
  JE Virus Nakayama Strain (≥2 to <5 yr; N = 9, 9) | 6.3 [5 to 40] | 27.2 [5 to 160]
  Wild Type Virus (≥2 to <5 yr; N = 9, 9) | 9.3 [5 to 40] | 17.1 [5 to 80]
  JE-CV Virus (≥9 mo to <2 yr; N = 13, 13) | 490.2 [40 to 5120] | 55.1 [5 to 320]
  JE Virus Nakayama (≥9 mo to <2 yr; N = 12, 13) | 5.3 [5 to 10] | 5.6 [5 to 10]
  Wild Type Virus (≥9 mo to <2 yr; N = 13, 13) | 136.3 [10 to 1280] | 17.0 [5 to 320]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from Day 14 to Day 42 (up to 28 days after completion of the course of vaccination).
Arm/Group | ChimeriVax™-JE | Mouse Brain Derived Vaccine
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 6/48 | 5/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ChimeriVax™-JE (N=48) | Mouse Brain Derived Vaccine (N=48)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (5)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications